CLINICAL TRIAL: NCT03421613
Title: A Double-Blind, Placebo-Controlled, Crossover Study to Evaluate the Efficacy and Tolerability of 3VM1001 Cream for the Treatment of Pain Associated With Post-Herpetic Neuralgia: A Proof of Concept Study
Brief Title: 3VM1001 Cream for the Treatment of Pain Associated With Post Herpetic Neuralgia (PHN)
Acronym: PHN
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: CDA Research Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3VM0416
Record Dates: First submitted 2018-01-30; First posted 2018-02-05 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-01

CONDITIONS: Treatment of PHN
Keywords: PHN, acute, herpes zoster
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster

STUDY DESIGN:
Intervention Model Description: Double-blind, Placebo-controlled, Crossover study to evaluate treatment and tolerability of the experimental product for treatment of post herpetic pain.
Who Masked: Participant, Care Provider
Masking Description: Subjects will be randomized to receive either treatment wih 3VM1001 cream or the comparator daily for 10 days followed by 5 day wash out period before 10 days of treatment with the comparator or investigational treatment, .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 3VM1001 cream (Experimental): Patients will be randomized to self treat with 2 g of VM1001 cream times daily for ten days, have a five day wash out period and then 10 days of self treatment with the comparator.
  Interventions: Drug: 3VM1001
- Placebo (Placebo Comparator): Patients will be randomized to self treat with either active product or placebo comparator thrice daily for 10 days followed by a 5 day wash out period then 10 days of experimental treatment thrice daily for 20 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 3VM1001 — Self treatment 3 times daily for 10 days
  Arms: 3VM1001 cream
Other: Placebo — Cream without investigational drug. Self treatment 3 times daily for 10 days
  Arms: Placebo

SUMMARY:
Post-herpetic neuralgia (PHN) is pain following acute herpes zoster; defined as pain lasting longer than 3 months. Current first line management consists of tricyclic anti-depressants and anti-convulsants such as gabapentin and pregabalin. There is an unmet medical need for treatments got topical therapies that demonstrate efficacy without serious side effects.

DETAILED DESCRIPTION:
Post-herpetic neuralgia (PHN) is defined as pain following acute herpes zoster (AHZ) lasting >3 months. PHN develops in about 10% of patients following an episode of AHZ. 95% of adults ate seropositive for varicella zoster virus antibodies, and are, therefore, at risk for AHZ and PHN. Wider use of AHZ vaccine approved in 2006 may reduce the incidence of PHN. Nevertheless, PHN may be severe and frequently interferes with daily activities and with sleep.

First line management of PHN pain currently is tricyclic anti-depressants and anti-convulsants such as gabapentin and pregabalin, and use of a 5% lidocaine patch. second line therapies include opioid analgesia and topical capsaicin: combinations of topical and systemic therapies may be used as well. These therapies have common side effects of dry mouth, constipation, sedation, urinary retention, nausea, somnolence, dizziness, weight gain and peripheral edema.

there is an unmet medial need for topical therapies that demonstrate efficacy without the significant side effects o the therapies mentioned above. 3VM cream, a low concentration of copper in a cream vehicle may b such a therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PHN for >3 months;
* Persistent pain for more than 6 months from appearance of herpes zoster rash that is not located above the scalp hairline, or in immediate proximity to mucous membranes (given the low toxicity of copper, PHN affecting the face and neck will be included, but subjects will be trained on avoidance of contact with the eyes or mouth);
* Age 18 years or older;
* Males or females of non-childbearing potential (i.e., 12 months or more of spontaneous amenorrhea, bilateral oophorectomy at least 6 months prior to randomization, hysterectomy with bilateral oophorectomy at least 6 months prior to randomization, or for females over 50 years of age, hysterectomy without bilateral oophorectomy at least 6 months prior to randomization); female subjects of childbearing potential must agree to use contraception (abstinence, birth control pills, rings or patches, diaphragm and spermicide, intrauterine device, condom and vaginal spermicide, surgical sterilization, vasectomy, progestin implant or injection); female partners of childbearing potential of male subjects must agree to use contraception as defined above;
* Persistent neuropathic pain that involves at least 1 dermatome and covering no more than 400 cm2 (the target area);
* Pain intensity in the target area of > 40mm on a 100mm VAS at screening;
* Intact skin over the target area to be treated;
* Subject agrees to take only the protocol-defined rescue medication as prescribed;
* All concurrent medications taken for any reason except for the treatment of PHN must be stable (dose, frequency) for 14 days;
* Ability to follow protocol with reference to cognitive and situational factors (eg. stable housing, ability to attend visits);
* Ability to read and write English;
* Ability to apply cream without assistance;
* Able to provide written informed consent.

Exclusion Criteria:

* Subject with systemic disease that would put him/her at an additional risk or limit his/her ability to participate in the study in the opinion of the investigator;
* Subject with known history of human immunodeficiency virus, hepatitis C, or hepatitis B;
* Malignancy other than basal cell carcinoma and carcinoma in situ within the past 2 years;
* Subject who has an active history of alcohol or drug abuse;
* Wilson's disease or other known disorder of copper metabolism;
* Known hypersensitivity or allergy to any component of the product, or to acetaminophen
* Pregnant and breastfeeding women.
* Subject with active herpes zoster lesions;
* Subject with open skin lesions or skin infections in the target area, or conditions over the target area such as eczema or psoriasis;
* Mild pain in the target area, characterized by VAS score of < 40 mm
* Pain in any other part of the body that could interfere with the patient's assessment of pain in the target area
* Subject who has taken concomitant medications for the treatment of PHN (except acetaminophen or gabapentin) in the last four weeks. If taking gabapentin the dose must have been stable for at least four weeks;
* Treatment with local anesthetic or steroids (including lidocaine patch, transcutaneous electrical nerve stimulation, etc.) in the last 2 weeks or nerve blocks within the last 30 days;
* Subject who has used capsaicin preparations on a regular basis in the 90 days prior to screening and at all in the past two weeks;
* Use of prohibited concomitant medications/therapies;

  1. Devices or therapeutic treatments for pain apart from acetaminophen as a rescue medication
  2. Systemic corticosteroids
  3. Other Investigational Drugs
  4. Chemotherapeutic drugs
  5. Immunotherapy
  6. Topical products applied to the target skin area
* Subject with history of serious mental illness or psychiatric illness such as dementia, depression, or schizophrenia, that will limit his/her ability to comply with study procedures;
* Subject who is unable to apply, or have a care giver apply, study ointment to the area of most painful skin segments, three times daily, once within 2 hours of waking, once mid-afternoon, and once prior to bedtime;
* Subject who has participated in any other investigational study within 60 days prior to screening;
* Subject who is employed by the Sponsor, study staff, and their families; or
* Subject who has any condition that would make him/her, in the opinion of the investigator or Sponsor, unsuitable for the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
The time averaged mean in a standard 100 mm visual analog scale (VAS). | 25 days total
  The time averaged mean of all patient pain scores over each study period; trend over time for each treatment sill be assessed by day of therapy to evaluate any increase or decrease in effect for each study treatment.

SECONDARY OUTCOMES:
Adverse Events, serious adverse events, and study discontinuation | 25 days total
  Collection of adverse events and the number of subjects discontinuing he study
Patient Global Expression of change Scale (PGIC) from baseline (day 0) to the end of each study period. | 25 days total
  This measure is a single-item rating by participants of their improvement with treatment on a 7-point sale that ranges from "very much improved" to very much worse" with "no change "the mid-midpoint".
Change in Patient Global Assessment of Treatment Satisfaction from baseline to the end of each study phase. | 25 days total
  Patient Global Assessment of Treatment Satisfaction from baseline to the end of each study phase. Patients will rate their overall satisfaction with study treatment using a 5-point categorical scale.
Use of Rescue medication | 25 days total
  recording of the use of rescue mediation at each phase of the study.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Medex Healthcare Research, Inc., Chicago, Illinois
  - Medex Healthcare Reasearch, Inc., New York, New York

IPD SHARING:
Plan to Share IPD: No